CLINICAL TRIAL: NCT02294968
Title: The Family Startup Program. A Randomized Controlled Trial of a Universal Group-based Parenting Support Program
Acronym: FIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Aarhus Kommune (Other); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIV1
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: First-time Pregnant Women and Their Partners

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Family Startup (Experimental): Family Startup plus usual pre- and postnatal care
  Interventions: Other: Family Startup (in Danish: Familieiværksætterne)
- Control (No Intervention): Usual pre- and postnatal care

INTERVENTIONS:
Other: Family Startup (in Danish: Familieiværksætterne) — Manualized parenting support program; see Center for Socialt Ansvar (2013)
  Arms: Family Startup

SUMMARY:
The aims of this study are to determine whether a group-based parent support program ("Family Startup") can lead to early improved parental sense of competence, family relations, and child development. Evaluation is based on a randomized controlled trial, with half of the participants receiving Family Startup and the other half receiving treatment as usual.

DETAILED DESCRIPTION:
Some knowledge exists about effectiveness of high-intensity delivery of parenting support to subsets of at risk families. To the best of our knowledge, however, little is known about effects of universal primary prevention programs.

The Family Startup Program is a structured format for implementing pre- and postnatal parenting support groups that prepare new families for their roles as parents as well as focus on enhancing parents' social network. The Family Startup Program gathers couples in groups and introduces participants to informal sources of support (e.g. by meeting and interacting with other new families) and to a broad range of community resources (e.g. financial advisers, child dentist, local solicitors, family counselors) providing them with information and parenting skills. The program content includes handling family finance, choice of paternity leave, couple communication, breastfeeding, network formation, ensuring dental health, sensitivity toward child signals, child rearing discipline, help-seeking behavior, home safety, and more.

A second formulated rational behind the program is that strengthening father involvement, social network formation and access to family services will serve to enhance family relationships, including parenting, coparenting and couple relationship quality. Through participation in Family Startup, families receive a long term connection with a health visitor in the community and are introduced to a broad range of community services. This can be expected to benefit optimal health service utility and ease access to resources for families and children with need. Improved child outcome are the ultimate goal. No scientific evaluation of program effects of the Family Startup program on child or family outcome was previously conducted.

ELIGIBILITY:
Inclusion Criteria:

-Parents, mothers as well as their partners, expecting their first child in the municipality of Aarhus are eligible for the study. This is because of the universal nature of the original program. Mothers are included if interested regardless of the fathers' decline. Biological fathers, registered partners, as well as non-registered partners are eligible.

Exclusion Criteria:

* Parents are excluded from the study if they are under the age of 18 years
* Not capable of managing own legal affairs
* Choose not to accept any routine pregnancy scans. These exclusion criteria are chosen to secure that study participants are legally responsible and that we are able to recruit them via the Department of Obstetrics and Gynaecology in connection with the nuchal translucency scan around week 12
* The father or partner is not included if the mother declines participation. The mother can choose to attend the Family Startup Program with a friend (i.e. a sister, friend or neighbor) but friends are not eligible for the study
* Finally, individuals are excluded if they are not able to understand the Danish oral presentation of the study information and hence cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1719 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
The Parenting Sense of Competence scale (PSOC) | measured when child is 9 months

SECONDARY OUTCOMES:
The Parenting Sense of Competence scale (PSOC) | measured when child is 18 months
Parenting Stress Scale | measured when child is 9 months
Breastfeeding duration | Duration before child is 9 months
Couple Satisfaction Index | measured when child is 9 months
Coparenting Relationship Scale | measured when child is 9 months

OTHER OUTCOMES:
number of visits to the general practitioner | measured when child is 9 months
Ages and Stages Questionnaire | measured when child is 9 months
School starting age | Before child is 8 years old

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Simonsen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Trillingsgaard TL, Maimburg RD, Simonsen M. Group-based parent support during the transition to parenthood: Primary outcomes from a randomised controlled trial. Soc Sci Med. 2021 Oct;287:114340. doi: 10.1016/j.socscimed.2021.114340. Epub 2021 Aug 30. PMID 34509031
- [Derived] Trillingsgaard T, Maimburg RD, Simonsen M. The Family Startup Program: study protocol for a randomized controlled trial of a universal group-based parenting support program. BMC Public Health. 2015 Apr 21;15:409. doi: 10.1186/s12889-015-1732-3. PMID 25895494